CLINICAL TRIAL: NCT02056769
Title: CT Perfusion Imaging to Predict Vasospasm in Subarachnoid Hemorrhage
Acronym: CT-PIPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-PIPS
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Subarachnoid Hemorrhage; Delayed Cerebral Ischemia; Cerebral Vasospasm; CT Perfusion
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT Perfusion (Experimental): All patients enrolled in the study
  Interventions: Radiation: CT Perfusion

INTERVENTIONS:
Radiation: CT Perfusion — Quantitative CT Perfusion imaging

SUMMARY:
Patients with brain hemorrhage resulting from a ruptured aneurysm (SAH) are at risk of developing a condition called vasospasm, one or two weeks after their hemorrhage. This is a major cause of stroke and death following SAH. A special type of CT scan, called CT perfusion, analyzes regional blood flow in the brain. We hypothesize that CT perfusion scans performed on admission and day 6 post-hemorrhage will enable us to predict which patients will go on to develop vasospasm.

DETAILED DESCRIPTION:
Rupture of a brain aneurysm results in a type of bleeding into the brain called subarachnoid hemorrhage (SAH). This is a substantial cause of morbidity and mortality world-wide: even with the best possible care, up to half of patients die and many are left disabled. Sometimes this is because the immediate brain damage from the bleed is very severe. However, many patients who seem to be doing well at first go on to develop something called "vasospasm": narrowing of large arteries in the brain. This results in the brain not getting enough blood, and the patient can suffer a stroke as a result. The lack of blood to the brain is called delayed cerebral ischemia (DCI), and is the major secondary cause of stroke and death in patients who survived the initial aneurysm rupture.

Vasospasm can be seen on angiograms (blood vessel imaging) in about two-thirds of SAH patients, and causes neurological symptoms of DCI in half of those patients. It usually develops about a week or so after SAH. Early diagnosis and treatment of cerebral vasospasm and delayed cerebral ischemia (DCI) reduces morbidity and mortality in SAH patients.

CT perfusion imaging is able to identify areas of reduced cerebral blood flow that are at risk of DCI and stroke. This technique is able to measure cerebral blood flow and blood volume (CBF, CBV), and calculates two other measures of cerebral perfusion: time to peak intensity (TTP) and mean transit time (MTT). Taken together, these provide information about the amount of blood the brain is receiving and whether the brain is compensating for any reduction in flow. This is helpful because seeing vasospasm on imaging is not enough to predict brain ischemia and stroke; the additional physiological information provided by the perfusion assessment strengthens the diagnosis of DCI. Early evidence suggests that CT perfusion is a fast, accurate, inexpensive and non-invasive method of brain imaging to identify patients with DCI after SAH, and guide appropriate therapy.

If we were able to successfully predict which patients are at high risk of DCI and/or stroke, we could intervene early. This could improve patient outcomes, while potentially allowing better use of limited intensive care and nursing resources. Other studies have shown that patients with DCI had altered perfusion prior to developing clinical symptoms, but we do not know whether we can use CT perfusion to predict patients at risk, or which CT perfusion measurements (e.g., CBF or TTP) are most useful.

The radiation risk associated with CT perfusion imaging is negligible, due to advances in CT technology which allow for routine simultaneous CT perfusion and CT angiogram (CTA) without a significant increase in radiation dose over conventional head CT-CTA alone. Judicious use of CT perfusion, through a structured algorithm that includes routine perfusion scans at admission and during the peak risk period for vasospasm, may actually decrease cumulative radiation dose for patients with SAH, by ruling out perfusion deficit and brain ischemia as a cause of decreased neurological function and limiting repeated angiograms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age (inclusive).
* Patient has a documented aneurysmal SAH.
* Patient or next of kin or person with appropriate power of attorney has provided written informed consent.
* Patient is willing and available for study follow-up visits.
* Patient has not been previously entered into this study.

Exclusion Criteria:

* Inability to obtain informed written consent.
* Patient is < 18 or > 75 years old.
* Patient is not expected to survive >24 hours (e.g. those presenting with loss of brain stem reflexes, or patients transferred to the Halifax Infirmary ICU for consideration of organ donation rather than active treatment)
* Patient history indicates high risk of non-compliance (e.g., substance abuse, psychosocial issues, etc.)
* Patient is currently breast feeding, or pregnant
* Patient is currently enrolled in another clinical study (device or drug).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
CBF Admit | Baseline
  Cerebral blood flow as measured on CT perfusion study on admission
CBV Admit | Baseline
  Cerebral blood volume as measured on CT perfusion study on admission
MTT Admit | Baseline
  Mean transit time as measured on CT perfusion study on admission
TTP Admit | Baseline
  Time to peak as measured on CT perfusion study on admission
CBF day 6 | Day 6 post-SAH
  Cerebral blood flow as measured on CT perfusion study on day 6 following subarachnoid hemorrhage
CBV day 6 | Day 6 post-SAH
  Cerebral blood volume as measured on CT perfusion study on day 6 following subarachnoid hemorrhage
MTT day 6 | Day 6 post-SAH
  Mean transit time as measured on CT perfusion study on day 6 following subarachnoid hemorrhage
TTP day 6 | Day 6 post-SAH
  Time to peak as measured on CT perfusion study on day 6 following subarachnoid hemorrhage

SECONDARY OUTCOMES:
Radiation Dose | 30 days post-SAH
  Total cumulative radiation dose from cranial imaging (CT Head, CT angiogram, CT perfusion, catheter angiography, endovascular coiling) during the initial hospital admission for SAH, up to 30 days post-SAH.

OTHER OUTCOMES:
Delayed Cerebral Ischemia | 30 days post-SAH
  Delayed cerebral ischemia is defined using a consensus recently agreed upon by an international panel of experts: namely, 1) stroke seen on CT or MRI scan, or proven at autopsy (not including stroke related to the aneurysm treatment), or 2) clinical deterioration presumed to be caused by DCI after other causes are excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Gwynedd E Pickett, MD, Principal Investigator — Capital District Health Authority, Halifax, Canada
Locations (1):
- Halifax Infirmary, Capital District Health Authority, Halifax, Nova Scotia, Canada